CLINICAL TRIAL: NCT00114725
Title: Laser-Assisted Versus Conventional Intracytoplasmic Sperm Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shady Grove Fertility Reproductive Science Center (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: P2004-1
Record Dates: First submitted 2005-06-16; First posted 2005-06-17 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2005-06

CONDITIONS: Infertility; Infertility, Male
Keywords: In Vitro Fertilization; Intracytoplasmic Sperm Injection; Oocytes; Zona Pellucida; Oolemma; Fertilization; Preimplantation Embryo Development
MeSH Terms: conditions — Infertility; Infertility, Male

INTERVENTIONS:
Procedure: Laser-assisted intracytoplasmic sperm injection

SUMMARY:
Laser-assisted intracytoplasmic sperm injection (ICSI) has been suggested as a more effective alterative to conventional ICSI when this method of insemination is indicated for patients undergoing in vitro fertilization (IVF). Laser-assisted ICSI differs from conventional ICSI in that a laser is used to drill a small hole through the hard outer coating surrounding an egg before the injection needle containing a single sperm is inserted into the egg. The hole eliminates compression of the egg that normally occurs with conventional ICSI, and thus may reduce the chance of damage. Laser-assisted ICSI is hypothesized to result in increased egg survival, and perhaps improved embryo quality, compared to conventional ICSI.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of infertility
* Scheduled for IVF with ICSI

Exclusion Criteria:

* Retrieval of fewer than 6 mature oocytes

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60
Dates: Start 2004-03; Study Completion 2004-10

PRIMARY OUTCOMES:
oocyte survival rate 1 day after ICSI

SECONDARY OUTCOMES:
normal fertilization rate 1 day after ICSI
embryo cell numbers 2 and 3 days after ICSI
embryo fragmentation rates 2 and 3 days after ICSI
embryo compaction rate through day 7 after ICSI
blastocyst formation rate through day 7 after ICSI

CONTACTS AND LOCATIONS:
Overall Officials: Alana Davis, BS, Principal Investigator — Shady Grove Fertility Reproductive Science Center; Kevin S Richter, PhD, Study Director — Shady Grove Fertility Reproductive Science Center
Locations (1):
- Shady Grove Fertility Reproductive Science Center, Rockville, Maryland, United States

REFERENCES:
- [Background] Mikhailusov SV, Bart BIa, Siluianov SV, Mikhailusova MP, Nikolaeva AS. [Duodenogastric reflux and gastric pathology in the elderly patients]. Eksp Klin Gastroenterol. 2010;(12):54-9. Russian. PMID 21560622
- [Background] Kurashige H, Cateau H. Dendritic slow dynamics enables localized cortical activity to switch between mobile and immobile modes with noisy background input. PLoS One. 2011;6(9):e24007. doi: 10.1371/journal.pone.0024007. Epub 2011 Sep 8. PMID 21931635
- [Background] Chand AL, Wijayakumara DD, Knower KC, Herridge KA, Howard TL, Lazarus KA, Clyne CD. The orphan nuclear receptor LRH-1 and ERalpha activate GREB1 expression to induce breast cancer cell proliferation. PLoS One. 2012;7(2):e31593. doi: 10.1371/journal.pone.0031593. Epub 2012 Feb 16. PMID 22359603
- [Background] Semiglazov VF, Paltuev RM, Remizov AS, Semiglazov VV, Dashian GA, Bessonov AA, Pen'kov KD, Vasil'ev AG, Semiglazova TIu, Kolar'kova VV. [The role of nanotechnology in creating novel antitumor agents]. Vopr Onkol. 2011;57(5):636-40. Russian. PMID 22238935
- [Background] Rienzi L, Ubaldi F, Martinez F, Minasi MG, Iacobelli M, Ferrero S, Tesarik J, Greco E. Clinical application of laser-assisted ICSI: a pilot study. Eur J Obstet Gynecol Reprod Biol. 2004 Jul 1;115 Suppl 1:S77-9. doi: 10.1016/j.ejogrb.2004.01.017. PMID 15196721